CLINICAL TRIAL: NCT04715906
Title: Coping Options for Parent Empowerment
Brief Title: Project COPE (Coping Options for Parent Empowerment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, Assistant Chair for Academic Affairs and Research, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20201530
Record Dates: First submitted 2020-12-29; First posted 2021-01-20 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UP-Caregiver Group (Experimental): Unified Protocol (UP) Caregiver Group will receive the UP for Transdiagnostic Treatment of Emotional Disorders for Caregivers intervention via telehealth using Zoom for a minimum of 4 up to 8 sessions ideally within 8 weeks.
  Interventions: Behavioral: UP-Caregiver

INTERVENTIONS:
Behavioral: UP-Caregiver — The Unified Protocol (UP) is a telehealth group session using Zoom with each session lasting approximately 60-90 minutes. The sessions will focus on a variety of Cognitive Behavior Therapy techniques. These sessions may include teaching coping skills, goal setting, parent-child problem solving and communication, and motivation during this pandemic.

SUMMARY:
The purpose of this research study is to collect information to better understand caregiver responses to COVID-19 stress and to help caregivers of children with Autism Spectrum Disorder (ASD) cope with these stressors.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to consent to participate via RedCap
2. Indicate a mild or greater elevation on screening measures of anxiety and/or depression
3. Not meet any exclusion criteria.
4. Lives in Florida
5. Has a child between the ages of 4-13 years who has been diagnosed with ASD
6. Speaks either English or Spanish primarily
7. Has technical capacity to participate in Zoom sessions on a mobile device or preferably a computer

Exclusion Criteria:

1. Severe mental illness (e.g., bipolar disorder, schizophrenia, an intellectual disability, psychosis, alcohol use disorder, substance use disorder) or hospitalization for mental health concerns or suicide attempt. Parents may receive concurrent psychiatric or psychological intervention services but may be excluded if the severity of current mental illness is such that outpatient, weekly group treatment would be considered inappropriate.
2. Parents who report any prior arrest for child endangerment, child abuse or child neglect may also be excluded.
3. Parents who have Moderate or greater risk of suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety levels as measured by GAD-7 | Baseline, 6 Weeks
  Parent Psychopathology levels will be reported as the change in the Generalized Anxiety Disorder 7-item (GAD-7) scores. GAD-7 is a 7-item measure assessing the presence and severity of symptoms of anxiety. The Scale has a total score ranging from 0 to 21 with the higher scores indicating greater anxiety.
Change in depressive symptoms as measured by the PHQ | Baseline, 6 Weeks
  Parent Psychopathology levels will be reported as the change in the Patient Health Questionnaire (PHQ) scores. PHQ is a 9-item measure assessing the severity of depressive symptoms. It has a total score ranging from 0 to 27 with the higher scores indicating greater depressive symptoms.

SECONDARY OUTCOMES:
Change in parenting beliefs as measured by the PSOC Scale | Baseline, 6 Weeks
  Parenting Sense of Competence (PSOC) scale is a 17-item measure of parenting self-efficacy and satisfaction. It has a total score ranging from 17 to 102 with the higher scores indicating greater self-efficacy and satisfaction in the parenting role.
Change in Hope as measured by the State Hope Scale | Baseline, 6 Weeks
  State Hope Scale is a 6-item measure designed to evaluate hope in adults. It has a total score ranging from 6 to 48 with the higher scores representing higher hope levels.
Acceptability of Intervention as measured by the Program Feedback Scale | 6 Weeks
  The Program Feedback Scale has a total score ranging from 0 to 28 with the higher score indicating perceived acceptability and feasibility of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No